CLINICAL TRIAL: NCT00736489
Title: A Phase II, Double-blind, Placebo-controlled, Randomised, 6-way Cross-over, Single-dose Study to Investigate the Local and Systemic Effects of 3 Doses of Inhaled AZD3199 (a β2-agonist) Compared to Formoterol in Asthmatic Patients
Brief Title: Single-dose Crossover Study to Investigate Pharmacodynamics of AZD3199
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D0570C00007; ToBe
Record Dates: First submitted 2008-08-15; First posted 2008-08-18 (Estimated); Results first posted 2014-04-03 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-04

CONDITIONS: Asthma; Airway Obstruction
Keywords: Asthma; airway obstruction; beta2-agonist; efficacy; inhalation
MeSH Terms: conditions — Asthma; Airway Obstruction; Respiratory Aspiration | interventions — AZD-3199; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- crossover dose 1 (Experimental): AZD3199 120 microgram
  Interventions: Drug: AZD3199
- crossover dose 2 (Experimental): AZD3199 480 microgram
  Interventions: Drug: AZD3199
- crossover dose 3 (Experimental): AZD3199 1920 microgram
  Interventions: Drug: AZD3199
- crossover dose 4 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- crossover dose 5 (Active Comparator): Formoterol 9 microgram
  Interventions: Drug: Formoterol
- crossover dose 6 (Active Comparator): Formoterol 36 microgram
  Interventions: Drug: Formoterol

INTERVENTIONS:
Drug: AZD3199 — Dry powder for inhalation, single dose
  Arms: crossover dose 1; crossover dose 2; crossover dose 3
Drug: Formoterol — Dry powder for inhalation, single dose
  Other Names: Oxis
  Arms: crossover dose 5; crossover dose 6
Drug: Placebo — Dry powder for inhalation, single dose
  Arms: crossover dose 4

SUMMARY:
The purpose of this study is to investigate the pharmacodynamics of single doses of AZD3199 in asthmatic patients.

ELIGIBILITY:
Inclusion Criteria:

* Asthmatic patients with pre-bronchodilatory FEV1 above 60% of predicted normal and above 1.5 liters.
* Men and post-menopausal women above 18 years of age.
* Reversible airway obstruction in response to classical beta2-agonist (salbutamol)
* Non/ex-smokers

Exclusion Criteria:

* Any clinically significant disease or disorder other than asthma
* Any clinically relevant abnormal findings at screening examinations
* Treatment with systemic glucocorticosteroids within the past 30 days
* Inhaled corticosteroid use if dosing is not kept constant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2008-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof Leif Bjermer, MD, PhD, Principal Investigator — University Hospital in Lund, Sweden
Locations (4):
- Research Site, Hvidovre, Denmark
- Sweden (3):
  - Research Site, Gothenburg
  - Research Site, Luleå
  - Research Site, Lund

REFERENCES:
- [Derived] Bjermer L, Rosenborg J, Bengtsson T, Lotvall J. Comparison of the bronchodilator and systemic effects of AZD3199, an inhaled ultra-long-acting beta(2)-adrenoceptor agonist, with formoterol in patients with asthma. Ther Adv Respir Dis. 2013 Oct;7(5):264-71. doi: 10.1177/1753465813497527. Epub 2013 Aug 1. PMID 23907810
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=238&filename=CSR-D0570C00007.pdf
- See also: D0570C00007 CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=238&filename=D0570C00007.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study has been performed in Sweden and Denmark at two University hospital clinics and two CROs. The recruitment period was between 11 August 2008 to 22 October 2008.
Groups:
- APCDEBa: AZD3199 120 Mcg followed by Placebo followed by AZD3199 1920 Mcg followed by Formoterol 9 Mcg followed by Formoterol 36 Mcg followed by AZD3199 480 Mcg.
- BADEPCa: AZD3199 480 Mcg followed by AZD3199 120 Mcg followed by Formoterol 9 Mcg followed by Formoterol 36 Mcg followed by Placebo followed by AZD3199 1920 Mcg.
- CBEPADa: AZD3199 1920 Mcg followed by AZD3199 480 Mcg followed by Formoterol 36 Mcg followed by Placebo followed by AZD3199 120 Mcg followed by Formoterol 9 Mcg .
- DCPABEa: Formoterol 9 Mcg followed by AZD3199 1920 Mcg followed by Placebo followed by AZD3199 120 Mcg followed by AZD3199 480 Mcg followed by Formoterol 36 Mcg.
- EDABCPa: Formoterol 36 Mcg followed by Formoterol 9 Mcg followed by AZD3199 120 Mcg followed by AZD3199 480 Mcg followed by AZD3199 1920 Mcg followed by Placebo.
- PEBCDAa: Placebo followed by Formoterol 36 Mcg followed by AZD3199 480 Mcg followed by AZD3199 1920 Mcg followed by Formoterol 9 Mcg followed by AZD3199 120 Mcg.
Period: Period 1
Arm/Group | APCDEBa | BADEPCa | CBEPADa | DCPABEa | EDABCPa | PEBCDAa
Started | 6 (Cross-over study) | 5 | 6 | 7 | 7 | 6
Completed | 5 | 5 | 6 | 7 | 7 | 5
Not Completed | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1
Period: Period 2
Arm/Group | APCDEBa | BADEPCa | CBEPADa | DCPABEa | EDABCPa | PEBCDAa
Started | 5 | 5 | 6 | 7 | 7 | 5
Completed | 5 | 5 | 6 | 7 | 7 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | APCDEBa | BADEPCa | CBEPADa | DCPABEa | EDABCPa | PEBCDAa
Started | 5 | 5 | 6 | 7 | 7 | 5
Completed | 5 | 5 | 6 | 7 | 7 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | APCDEBa | BADEPCa | CBEPADa | DCPABEa | EDABCPa | PEBCDAa
Started | 5 | 5 | 6 | 7 | 7 | 5
Completed | 5 | 5 | 6 | 7 | 7 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 5
Arm/Group | APCDEBa | BADEPCa | CBEPADa | DCPABEa | EDABCPa | PEBCDAa
Started | 5 | 5 | 6 | 7 | 7 | 5
Completed | 5 | 5 | 6 | 7 | 7 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 6
Arm/Group | APCDEBa | BADEPCa | CBEPADa | DCPABEa | EDABCPa | PEBCDAa
Started | 5 | 5 | 6 | 7 | 7 | 5
Completed | 5 | 5 | 6 | 7 | 7 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Baseline Total: Total number of patients randomized and treated in the study
Arm/Group | Baseline Total
Number analyzed (Participants) | 37
Age, Continuous [Mean (Full Range); unit: years] | 40.3 [22 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 32

OUTCOME MEASURES:

1. Primary Outcome: FEV1 Peak Effect Within 0 - 24 h Post-dose
Description: Maximum FEV1 value
Time Frame: 0, 5min, 15min, 30min, 1h, 2h, 4h, 6h, 8h, 10h, 12h, 14h, 18h, 22h, 24h
Population: Two patients discontinued after the first treatment period and were excluded from pharmacodynamic analysis set since these patients are non-informative regarding treatment differences. One patient on Placebo treatment had data not sufficient for computing PD parameters and for subsequent analysis.
Measure: Mean (Standard Deviation); unit: L
Groups:
- AZD3199 120 mcg: AZD3199 120 Mcg inhaled via Turbuhaler
- AZD3199 480 mcg: AZD3199 480 Mcg inhaled via Turbuhaler
- AZD3199 1920 mcg: AZD3199 1920 Mcg inhaled via Turbuhaler
- Formoterol 9 mcg: Formoterol 9 Mcg inhaled via Turbuhaler
- Formoterol 36 mcg: Formoterol 36 Mcg inhaled via Turbuhaler
- Placebo: Placebo inhaled via Turbuhaler
Arm/Group | AZD3199 120 mcg | AZD3199 480 mcg | AZD3199 1920 mcg | Formoterol 9 mcg | Formoterol 36 mcg | Placebo
Number analyzed (Participants) | 35 | 35 | 35 | 35 | 35 | 34
L | 3.56 (0.94) | 3.62 (0.94) | 3.70 (1.02) | 3.62 (1.01) | 3.69 (0.97) | 3.44 (0.99)

2. Primary Outcome: E22-26: the Average of the FEV1 Value Between 22 and 26 h Post Dose for Every Treatment Visit.
Description: Residual FEV1 24 h post-dose
Time Frame: 22- 26 h post dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | AZD3199 120 mcg | AZD3199 480 mcg | AZD3199 1920 mcg | Formoterol 9 mcg | Formoterol 36 mcg | Placebo
Number analyzed (Participants) | 35 | 35 | 35 | 35 | 35 | 34
L | 3.31 (0.96) | 3.35 (0.93) | 3.40 (0.94) | 3.26 (0.94) | 3.36 (0.97) | 3.23 (0.96)

3. Primary Outcome: S-potassium, Peak Effect Over 0 - 4 h Post-dose
Description: Minimum S-potassium concentration (A well-known effect of beta2-agonists (AZD3199 is a beta2-agonist) is a reduction in serum potassium levels. The minimum value has therefore been evaluated.
Time Frame: 0, 15min, 30min,1h, 2h, 4h
Population: Two patients discontinued after the first treatment period and were excluded from pharmacodynamic analysis set since these patients are non-informative regarding treatment differences. Two patients on AZD3199 1920 mcg had data not sufficient for computing PD parameters and for subsequent analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | AZD3199 120 mcg | AZD3199 480 mcg | AZD3199 1920 mcg | Formoterol 9 mcg | Formoterol 36 mcg | Placebo
Number analyzed (Participants) | 35 | 35 | 33 | 35 | 35 | 35
mmol/L | 4.04 (0.19) | 4.03 (0.25) | 3.98 (0.28) | 4.04 (0.20) | 3.84 (0.21) | 4.04 (0.23)

4. Primary Outcome: S-potassium, Average Effect Over 0 - 4 h Post-dose
Description: Average S-potassium concentration
Time Frame: 0, 15min, 30min,1h, 2h, 4h
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | AZD3199 120 mcg | AZD3199 480 mcg | AZD3199 1920 mcg | Formoterol 9 mcg | Formoterol 36 mcg | Placebo
Number analyzed (Participants) | 35 | 35 | 33 | 35 | 35 | 35
mmol/L | 4.22 (0.19) | 4.21 (0.26) | 4.17 (0.26) | 4.19 (0.20) | 3.99 (0.17) | 4.21 (0.25)

5. Secondary Outcome: FEV1 Effect at 5 Min Post-dose
Description: FEV1 at 5 minutes
Time Frame: 5min
Population: Two patients discontinued after the first treatment period and were excluded from pharmacodynamic analysis set since these patients are non-informative regarding treatment differences. Two patients on Placebo and 1 on AZD3199 480 mcg had data not sufficient for computing PD parameters and for subsequent analysis.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | AZD3199 120 mcg | AZD3199 480 mcg | AZD3199 1920 mcg | Formoterol 9 mcg | Formoterol 36 mcg | Placebo
Number analyzed (Participants) | 35 | 34 | 35 | 35 | 35 | 33
L | 3.36 (0.88) | 3.38 (0.92) | 3.33 (1.03) | 3.37 (0.95) | 3.47 (0.93) | 3.13 (0.86)

6. Secondary Outcome: FEV1 Average Effect Over 0 - 24 h Post-dose
Description: FEV1 average effect over 24 h dosing interval
Time Frame: 0, 5min, 15min, 30min, 1h, 2h, 4h, 6h, 8h, 10h, 12h, 14h, 18h, 22h, 24h
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | AZD3199 120 mcg | AZD3199 480 mcg | AZD3199 1920 mcg | Formoterol 9 mcg | Formoterol 36 mcg | Placebo
Number analyzed (Participants) | 35 | 35 | 35 | 35 | 35 | 34
L | 3.31 (0.93) | 3.36 (0.91) | 3.44 (0.95) | 3.35 (0.98) | 3.46 (0.96) | 3.19 (0.95)

7. Secondary Outcome: FEV1 Average Effect Over 0 - 12 h Post-dose
Description: FEV1 average effect over 12 h day-time period
Time Frame: 0, 5min, 15min, 30min, 1h, 2h, 4h, 6h, 8h, 10h, 12h
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | AZD3199 120 mcg | AZD3199 480 mcg | AZD3199 1920 mcg | Formoterol 9 mcg | Formoterol 36 mcg | Placebo
Number analyzed (Participants) | 35 | 35 | 35 | 35 | 35 | 34
L | 3.33 (0.92) | 3.40 (0.89) | 3.48 (0.97) | 3.40 (0.98) | 3.51 (0.95) | 3.20 (0.96)

8. Secondary Outcome: FEV1 Average Effect Over 12 - 24 h Post-dose
Description: FEV1 average effect over 12 h night-time period
Time Frame: 12h, 14h, 18h, 22h, 24h
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | AZD3199 120 mcg | AZD3199 480 mcg | AZD3199 1920 mcg | Formoterol 9 mcg | Formoterol 36 mcg | Placebo
Number analyzed (Participants) | 35 | 35 | 35 | 35 | 35 | 34
L | 3.28 (0.95) | 3.33 (0.92) | 3.41 (0.94) | 3.30 (0.98) | 3.40 (0.98) | 3.19 (0.95)

9. Secondary Outcome: Systolic Blood Pressure, Peak Effect Over 0 - 4 h Post-dose
Description: Maximum SBP value over 4 h
Time Frame: 0, 30min, 2h, 4h
Population: Two patients discontinued after the first treatment period and were excluded from pharmacodynamic analysis set since these patients are non-informative regarding treatment differences.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AZD3199 120 mcg | AZD3199 480 mcg | AZD3199 1920 mcg | Formoterol 9 mcg | Formoterol 36 mcg | Placebo
Number analyzed (Participants) | 35 | 35 | 35 | 35 | 35 | 35
mmHg | 126.8 (14.5) | 128.3 (13.4) | 127.4 (12.0) | 127.3 (13.2) | 129.9 (12.1) | 126.4 (14.4)

10. Secondary Outcome: Systolic Blood Pressure, Average Effect Over 0 - 4 h Post-dose
Description: Average SBP value over 4 h
Time Frame: 0, 30min, 2h, 4h
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AZD3199 120 mcg | AZD3199 480 mcg | AZD3199 1920 mcg | Formoterol 9 mcg | Formoterol 36 mcg | Placebo
Number analyzed (Participants) | 35 | 35 | 35 | 35 | 35 | 35
mmHg | 121.1 (13.7) | 121.8 (11.8) | 121.3 (11.9) | 120.9 (12.8) | 122.6 (11.8) | 121.3 (13.5)

11. Secondary Outcome: Diastolic Blood Pressure, Peak Effect Over 0 - 4 h Post-dose
Description: Minimum DBP value over 4 h
Time Frame: 0, 30min, 2h, 4h
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AZD3199 120 mcg | AZD3199 480 mcg | AZD3199 1920 mcg | Formoterol 9 mcg | Formoterol 36 mcg | Placebo
Number analyzed (Participants) | 35 | 35 | 35 | 35 | 35 | 35
mmHg | 67.3 (10.3) | 67.6 (7.9) | 66.7 (9.6) | 66.9 (9.1) | 66.7 (9.6) | 68.8 (8.0)

12. Secondary Outcome: Diastolic Blood Pressure, Average Effect Over 0 - 4 h Post-dose
Description: Average DBP value over 4 h
Time Frame: 0, 30min, 2h, 4h
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AZD3199 120 mcg | AZD3199 480 mcg | AZD3199 1920 mcg | Formoterol 9 mcg | Formoterol 36 mcg | Placebo
Number analyzed (Participants) | 35 | 35 | 35 | 35 | 35 | 35
mmHg | 71.4 (10.0) | 72.0 (8.9) | 71.6 (9.5) | 71.5 (9.2) | 71.0 (8.6) | 72.7 (8.4)

13. Secondary Outcome: Pulse, Peak Effect Over 0 - 4 h Post-dose
Description: Maximum pulse over 4 h
Time Frame: 0, 30min, 2h, 4h
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | AZD3199 120 mcg | AZD3199 480 mcg | AZD3199 1920 mcg | Formoterol 9 mcg | Formoterol 36 mcg | Placebo
Number analyzed (Participants) | 35 | 35 | 35 | 35 | 35 | 35
bpm | 62.1 (9.4) | 65.0 (11.0) | 66.7 (9.9) | 63.6 (11.0) | 67.3 (11.6) | 65.3 (10.4)

14. Secondary Outcome: Pulse, Average Effect Over 0 - 4 h Post-dose
Description: Average pulse over 4 h
Time Frame: 0, 30min, 2h, 4h
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | AZD3199 120 mcg | AZD3199 480 mcg | AZD3199 1920 mcg | Formoterol 9 mcg | Formoterol 36 mcg | Placebo
Number analyzed (Participants) | 35 | 35 | 35 | 35 | 35 | 35
bpm | 57.1 (8.0) | 59.0 (8.7) | 61.9 (9.1) | 58.6 (9.4) | 62.8 (10.1) | 58.8 (8.8)

15. Secondary Outcome: Heart Rate, Peak Effect Over 0 - 4 h Post-dose
Description: Maximum heart rate over 4 h
Time Frame: 0, 30min, 2h, 4h
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | AZD3199 120 mcg | AZD3199 480 mcg | AZD3199 1920 mcg | Formoterol 9 mcg | Formoterol 36 mcg | Placebo
Number analyzed (Participants) | 35 | 35 | 35 | 35 | 35 | 35
bpm | 64.0 (8.8) | 64.1 (9.6) | 66.9 (9.5) | 63.8 (10.2) | 66.8 (10.9) | 64.5 (11.3)

16. Secondary Outcome: Heart Rate, Average Effect Over 0 - 4 h Post-dose
Description: Average heart rate over 4 h
Time Frame: 0, 30min, 2h, 4h
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | AZD3199 120 mcg | AZD3199 480 mcg | AZD3199 1920 mcg | Formoterol 9 mcg | Formoterol 36 mcg | Placebo
Number analyzed (Participants) | 35 | 35 | 35 | 35 | 35 | 35
bpm | 58.3 (7.9) | 59.0 (8.5) | 61.8 (9.0) | 58.6 (9.2) | 62.7 (10.0) | 58.1 (8.6)

17. Secondary Outcome: QTcB, Peak Effect Over 0 - 4 h Post-dose
Description: Maximum QTc Bazett over 4 h
Time Frame: 0, 30min, 2h, 4h
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | AZD3199 120 mcg | AZD3199 480 mcg | AZD3199 1920 mcg | Formoterol 9 mcg | Formoterol 36 mcg | Placebo
Number analyzed (Participants) | 35 | 35 | 35 | 35 | 35 | 35
ms | 412 (21.6) | 407 (22.8) | 413 (22.0) | 408 (21.6) | 415 (24.6) | 408 (20.8)

18. Secondary Outcome: QTcB, Average Effect Over 0 - 4 h Post-dose
Description: Average QTc Bazett over 4 h
Time Frame: 0, 30min, 2h, 4h
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | AZD3199 120 mcg | AZD3199 480 mcg | AZD3199 1920 mcg | Formoterol 9 mcg | Formoterol 36 mcg | Placebo
Number analyzed (Participants) | 35 | 35 | 35 | 35 | 35 | 35
ms | 398 (19.9) | 397 (22.3) | 402 (21.2) | 395 (21.4) | 406 (24.4) | 395 (19.8)

19. Secondary Outcome: Tremor, Peak Effect Over 0 - 4 h Post-dose
Description: Maximum tremor score (4 grade scale: 0=no, 1=mild, 2=moderate or 3=severe) over 4 h.
Time Frame: 0, 15min, 30min, 1h, 2h, 4h
Population: Two patients discontinued after the first treatment period and were excluded from pharmacodynamic analysis set since these patients are non-informative regarding treatment differences. One patient on Placebo, 1 patient on formoterol 36 mcg and 1 patient on AZD3199 480 mcg had no data for subsequent analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | AZD3199 120 mcg | AZD3199 480 mcg | AZD3199 1920 mcg | Formoterol 9 mcg | Formoterol 36 mcg | Placebo
Number analyzed (Participants) | 35 | 34 | 35 | 35 | 34 | 34
Score on a scale | 0.06 (0.24) | 0.06 (0.24) | 0.17 (0.45) | 0.11 (0.32) | 0.47 (0.66) | 0.03 (0.17)

20. Secondary Outcome: Tremor, Average Effect Over 0 - 4 h Post-dose
Description: Average tremor score (4 grade scale: 0=no, 1=mild, 2=moderate or 3=severe) over 4 h.
Time Frame: 0, 15min, 30min, 1h, 2h, 4h
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | AZD3199 120 mcg | AZD3199 480 mcg | AZD3199 1920 mcg | Formoterol 9 mcg | Formoterol 36 mcg | Placebo
Number analyzed (Participants) | 35 | 34 | 35 | 35 | 34 | 34
Score on a scale | 0.00 (0.02) | 0.02 (0.08) | 0.04 (0.11) | 0.05 (0.18) | 0.16 (0.34) | 0.01 (0.06)

21. Secondary Outcome: Palpitations, Peak Effect Over 0 - 4 h Post-dose
Description: Maximum palpitation score (4 grade scale: 0=no, 1=mild, 2=moderate or 3=severe) over 4 h
Time Frame: 0, 15min, 30min, 1h, 2h, 4h
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | AZD3199 120 mcg | AZD3199 480 mcg | AZD3199 1920 mcg | Formoterol 9 mcg | Formoterol 36 mcg | Placebo
Number analyzed (Participants) | 35 | 34 | 35 | 35 | 34 | 34
Score on a scale | 0.03 (0.17) | 0.03 (0.17) | 0.09 (0.37) | 0.00 (0.00) | 0.18 (0.52) | 0.00 (0.00)

22. Secondary Outcome: Palpitations, Average Effect Over 0 - 4 h Post-dose
Description: Average palpitation score (4 grade scale: 0=no, 1=mild, 2=moderate or 3=severe) over 4 h
Time Frame: 0, 15min, 30min, 1h, 2h, 4h
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | AZD3199 120 mcg | AZD3199 480 mcg | AZD3199 1920 mcg | Formoterol 9 mcg | Formoterol 36 mcg | Placebo
Number analyzed (Participants) | 35 | 34 | 35 | 35 | 34 | 34
Score on a scale | 0.00 (0.02) | 0.01 (0.05) | 0.02 (0.08) | 0.00 (0.00) | 0.11 (0.33) | 0.00 (0.00)

23. Secondary Outcome: Plasma AZD3199 Cmax
Description: Maximum plasma concentration of AZD3199 measured
Time Frame: 0, 5min, 15min, 30min, 1h, 2h, 4h, 8h, 12h, 24h
Population: Two patients discontinued after the first treatment period and were excluded from pharmacokinetic analysis set.
Measure: Geometric Mean (Full Range); unit: nmol/L
Arm/Group | AZD3199 120 mcg | AZD3199 480 mcg | AZD3199 1920 mcg | Formoterol 9 mcg | Formoterol 36 mcg | Placebo
Number analyzed (Participants) | 35 | 35 | 35 | 0 | 0 | 0
nmol/L | 0.99 [0.21 to 2.83] | 5.39 [1.32 to 12.4] | 24.55 [8.99 to 44.3] |  |  |

24. Secondary Outcome: Plasma AZD3199 AUC0-24
Description: Area under the plasma concentration curve from time 0 to 24 h post-dose
Time Frame: 0, 5min, 15min, 30min, 1h, 2h, 4h, 8h, 12h, 24h
Population: Two patients discontinued after the first treatment period and were excluded from pharmacokinetic analysis set.
Measure: Geometric Mean (Full Range); unit: nmol*h/L
Arm/Group | AZD3199 120 mcg | AZD3199 480 mcg | AZD3199 1920 mcg | Formoterol 9 mcg | Formoterol 36 mcg | Placebo
Number analyzed (Participants) | 35 | 35 | 35 | 0 | 0 | 0
nmol*h/L | 1.83 [0.3 to 5.2] | 9.75 [2.9 to 23.5] | 46.06 [14.6 to 106.2] |  |  |

ADVERSE EVENTS:
Arm/Group | AZD3199 120 mcg | AZD3199 480 mcg | AZD3199 1920 mcg | Formoterol 9 mcg | Formoterol 36 mcg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/35 | 0/35 | 0/35 | 0/35 | 0/36
Other Adverse Events (participants affected / at risk) | 4/36 | 3/35 | 10/35 | 2/35 | 4/35 | 6/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD3199 120 mcg (N=36) | AZD3199 480 mcg (N=35) | AZD3199 1920 mcg (N=35) | Formoterol 9 mcg (N=35) | Formoterol 36 mcg (N=35) | Placebo (N=36)
Headache (Nervous system disorders) | 1 | 3 | 4 | 2 | 3 | 2
Nasopharyngitis (Infections and infestations) | 3 | 1 | 4 | 0 | 1 | 4
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to any publication or disclosure, the PI provides AstraZeneca with preliminary data and drafts and with the proposed final manuscript. AstraZeneca shall have a period of 30 days from receipt of the proposed final manuscript to review it and may within such time frame require that submission for publication or disclosure be delayed.